CLINICAL TRIAL: NCT01920113
Title: A Comparison of Efficacy and Safety During Endoscopic Submucosal Dissection Between Dexmedetomidine-remifentanil and Propofol-remifentanil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2012-0621
Record Dates: First submitted 2013-07-23; First posted 2013-08-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Early Gastric Cancer Patients Who Were Scheduled for Endoscopic Submucosal Dissection
Keywords: Endoscopic submucosal dissection; propofol; remifentanil; dexmedetomidine; efficacy; safeness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DR group (Experimental): In Group DR, a bolus dose of 0.5mcg/kg dexmedetomidine was injected intravenously 5 minutes before the start of the procedure (Precedex®, Abbott, Istanbul, Turkey). And a continuous infusion dose of 0.3-0.7mcg/hr/kg was started.
  Interventions: Drug: Dexmedetomidine - remifentanil group
- PR group (Active Comparator): In Group PR, a bolus injection of 1 mg/kg of propofol was followed by a continuous infusion at a rate of 3-5mg/hr/kg(Pofol®, Dongkook Pharm. Co. Ltd., Seoul, Korea) using an infusion pump (Syringe Pump TE-331, Terumo Japan).
  Interventions: Drug: Propofol - remifentanil group

INTERVENTIONS:
Drug: Dexmedetomidine - remifentanil group
  Arms: DR group
Drug: Propofol - remifentanil group
  Arms: PR group

SUMMARY:
Adequate, safe sedation is essential for Endoscopic submucosal dissection. Dexmedetomidine is a potent and selective a2-adrenoceptor agonist used for sedative and analgesic effects, but it is limited to use alone. The investigators designed this study to compare the effect and safety of two sedatives, dexmedetomidine and propofol in Endoscopic Submucosal Dissection (ESD), when sufficient analgesia-remifentanil is administered all throughout the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20
* American Society of Anaesthesiologists(ASA) physical status classification I~III
* Early gastric cancer patients who were scheduled for Endoscopic submucosal dissection

Exclusion Criteria:

* Age < 20
* American Society of Anaesthesiologists(ASA) physical status classification IV
* those with end-organ diseases (i.e. heart failure, respiratory failure, hepatic failure, renal failure)
* known drug allergies or history of drug abuse
* psychological disease

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
A comparison of safety during endoscopic submucosal dissection between dexmedetomidine-remifentanil and propofol-remifentanil | right after the drugs had administered
  Safety : whether the complications as follows occur or not
  1. systolic blood pressure under 90mmHg or 20% out of range of the baseline SBP
  2. heart rate under 50bpm
  3. oxygen saturation under 90%, respiratory rate under 7 per minute

SECONDARY OUTCOMES:
A comparison of efficacy during endoscopic submucosal dissection between dexmedetomidine-remifentanil and propofol-remifentanil | right after the drugs had administered
  Efficacy :
  1. whether a bolus injection of 10 mg of propofol was administered or not
  2. evaluating the depth of sedation using MOAA/S scale all through the procedure
  3. whether the en bloc resection, complete resection were done or not under the sedation

OTHER OUTCOMES:
A comparison of patient's satisfaction during endoscopic submucosal dissection between dexmedetomidine-remifentanil and propofol-remifentanil | within 24hrs after procedure
  Patients' satisfaction : investigate in four steps questionaire (very good, good, bearable and unbearable) when the patients' were discharged from PACU
A comparison of gastric motility, easiness for procedure, operator's satisfaction during endoscopic submucosal dissection between dexmedetomidine-remifentanil and propofol-remifentanil | right after the drugs had administered
  Subjects' motility grading during procedure, easiness of procedure, operator's satisfaction : investigate in four steps questionaires by the operator after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology & Pain Medicine, Yonsei university college of medicine, Seoul, South Korea

REFERENCES:
- [Derived] Kim N, Yoo YC, Lee SK, Kim H, Ju HM, Min KT. Comparison of the efficacy and safety of sedation between dexmedetomidine-remifentanil and propofol-remifentanil during endoscopic submucosal dissection. World J Gastroenterol. 2015 Mar 28;21(12):3671-8. doi: 10.3748/wjg.v21.i12.3671. PMID 25834336